CLINICAL TRIAL: NCT05134467
Title: Prospective, Single-center, Observational Study on the Assessment of Process and Outcome of Protocol-based Weaning From Mechanical Ventilation in the Medical Patients
Brief Title: Assessment of Process and Outcome of Protocol-based Weaning From Mechanical Ventilation in the Medical Patients
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kyeongman Jeon, Professor of Medicine, Samsung Medical Center
Other Study IDs: SMC 2017-08-141-009
Record Dates: First submitted 2021-11-10; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Ventilator Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, single-center, observational study to describe characteristics of weaning process and factors associated with duration of weaning and its outcomes in all consecutive adult (aged 19 years and older) patients receiving mechanical ventilation for at least two calendar days in medical intensive care units since November 2017. Details of the patients' weaning process and spontaneous breathing trial (SBT) in addition to clinical, laboratory, and outcome data will be collected in a specified format on the day of the assessment by respiratory care practitioners.

DETAILED DESCRIPTION:
Study design and objectives: This is a prospective, single-center, observational study to address key issues relating to weaning from mechanical ventilation (MV) in medical intensive care units. This study aims to describe characteristics of weaning process and factors associated with duration of weaning and its outcomes.

Inclusion criteria: All consecutive adult (aged 19 years and older) patients receiving MV for at least two calendar days in medical intensive care units since November 2017 will be screened daily.

Exclusion criteria: None

Protocol based weaning process: Every morning, respiratory care practitioners assess a patient's readiness to be weaned from MV in all patients who received MV for more than 24 h. First, the patient's condition, including improvement of the underlying cause of respiratory failure, clinical stability, and adequacy of pulmonary function and oxygenation are comprehensively evaluated. If the patient fulfill all of the criteria of readiness for weaning trials, SBT is conducted according to the protocol to assess the ability of the patient for spontaneous breathing; if the patient does not fulfill the criteria, no further weaning process is performed on that day. Our hospital performed the T-piece trial, in which supplemental oxygen was provided through a T-piece connected to an endotracheal tube or tracheostomy tube, on all patients until July 2019. From July 2019, SBT has been performed with inspiratory pressure augmentation (the ventilator is set with a pressure support of 8 cmH2O and zero-positive end-expiratory pressure) for patients who received MV through an endotracheal tube according to the revised weaning protocol. Tolerance for SBT is evaluated for 30 min on the first attempt and for 2 h after the second attempt, regardless of the method used. However, if a sign of SBT failure is identified even before the target duration, the trial is immediately stopped. When the patient satisfies all the criteria for successful SBT, extubation is performed immediately, and supplemental oxygen is provided by a high-flow nasal cannula for at least 24 h in patients with an endotracheal tube; administration of supplemental oxygen is continued through a T-piece system in patients with tracheostomy. Decisions about when and how to perform a tracheostomy are left to the discretion of the clinicians and are not guided by a prescribed algorithm.

Data collection and clinical outcomes: Clinical, laboratory, and outcome data will be prospectively collected by a trained study coordinator. The demographics of the patients and major cause of intubation will be evaluated and recorded by the physicians on the day of MV support initiation. Details of the patients' weaning readiness and SBT will be recorded in a specified format on the day of the assessment by respiratory care practitioners. The values of the MV setting and respiratory parameters are synchronized to the hospital electronic medical chart and recorded every hour, and we will collect the values at 8 am on the day of the first SBT. Clinical outcomes will be assessed by the successful weaning defined according to Weaning Outcome according to a New Definition (WIND) study and WIND classification of weaning.

Ethical Approval and Patient Consent: The Institutional Review Board of Samsung Medical Center approved this study and waived the requirement for informed consent, because this study is pure observation and data collection program that involves no more than minimal risk, the data collected are part of routine clinical care that would not adversely affect rights and welfare of subject, and the data will be anonymized.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult patients receiving mechanical ventilation for at least two calendar days in medical intensive care units

Exclusion Criteria:

* None

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving mechanical ventilation for at least two calendar days in medical intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Successful weaning | 6 months from MV
  Extubation without death or reintubation within the next 7 days of spontaneous breathing trial or discharge from intensive care unit without invasive mechanical ventilation (MV) within 7 days, whichever comes first for intubated patients and as spontaneous ventilation through tracheostomy without any MV during 7 consecutive days or discharged with spontaneous breathing, whichever comes first for patients with tracheostomy after the first separation attempt
Weaning outcomes by the Weaning Outcome according to a New Definition (WIND) classification | 6 months from MV
  Group 1 (short weaning), the first attempt result in the termination of the weaning process within 1 day
  Group 2 (difficult weaning), the weaning process is completed after more than 1 day but in less than 1 week after the first separation attempt
  Group 3 (prolonged weaning), the weaning process is still not terminated 7 days after the first separation attempt.

CONTACTS AND LOCATIONS:
Overall Officials: Kyeongman Jeon, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Na SJ, Ko RE, Nam J, Ko MG, Jeon K. Factors associated with prolonged weaning from mechanical ventilation in medical patients. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221117005. doi: 10.1177/17534666221117005. PMID 35943272